CLINICAL TRIAL: NCT01541748
Title: Axis™ Allograft Dermis for Female Pelvic Floor Repair: a Prospective Post Market Study
Status: Completed | Type: Observational
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: CP009SU
Record Dates: First submitted 2012-02-17; First posted 2012-03-01 (Estimated); Results first posted 2020-06-18 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AXIS Allograft Dermis: Participants receiving AXIS Allograft Dermis for anterior, posterior or combined (anterior and posterior) female pelvic floor repair.
  Interventions: Other: Axis

INTERVENTIONS:
Other: Axis — Coloplast's Axis™ Allograft Dermis is used for anterior, posterior or combined (anterior and posterior) pelvic organ prolapse repair.

SUMMARY:
This study is a prospective, single arm, multi-center, post-market study to evaluate the efficacy of Axis™ Allograft Dermis used for anterior, posterior or combined (anterior and posterior) pelvic organ prolapse repair.

DETAILED DESCRIPTION:
The study population will be adult female patients with pelvic organ prolapse, POP-Q Stage ≥ 2 that are clinically indicated for surgical intervention with Axis Allograft Dermis in the anterior, posterior or combined (anterior and posterior) compartments.

ELIGIBILITY:
Inclusion Criteria:

* Adult female at least 18 years of age.
* Willing and able to provide written informed consent.
* Confirmed pelvic organ prolapse (POP) of Stage 2 or higher as determined by POP-Q prolapse grading requiring surgical intervention in the anterior, posterior or combined (anterior and posterior) compartment.
* Willing and able to complete all follow-up visits and procedures indicated in this protocol.

Exclusion Criteria:

* Concurrent surgical treatment of pelvic organ prolapse using anything other than the Axis Dermis.[Note: concurrent mid-urethral sling placement for treatment of stress urinary incontinence is allowed].
* Confirmed Stage 2 or higher prolapse as determined by POP-Q prolapse grading for a compartment that is not being repaired in the same procedure. (Concurrent POP-Q Stage 1 repair is at the physician's discretion.)
* Previous pelvic organ prolapse repair using biologic, or synthetic grafts. [Note: previous mid-urethral sling for treatment of stress urinary incontinence is allowed]
* Pregnant or a desire to become pregnant in the future.
* Previous radiation or other treatments for cancer in the pelvic area.
* Severe urogenital atrophy.
* Immunosuppression and/or current systemic steroid user.
* Any contraindication to the surgical procedure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be adult female patients with pelvic organ prolapse, POP-Q Stage ≥ 2 that are clinically indicated for surgical intervention with Axis human tissue in the anterior, posterior, or combined (anterior and posterior) compartments at the institutions designated for this study.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2011-11; Primary Completion 2018-11-11 (Actual); Study Completion 2018-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Whitmore, MD, Principal Investigator — Virtua Female Pelvic Medicine
Locations (5):
- United States (5):
  - Cleveland Clinic Florida, Weston, Florida
  - Boston Urogynecology Associates, Cambridge, Massachusetts
  - Female Pelvic Medicine and Urogynecology Institute of MI/Grand Rapids Women's Health, Grand Rapids, Michigan
  - The Institute for Female Pelvic Medicine and Reconstructive Surgery, Allentown, Pennsylvania
  - Philadelphia Urosurgical Associates, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Seventy-four subjects were consented. Five subjects did not meet inclusion/exclusion criteria and one subject was not implanted with a study device.
Groups:
- Axis Allograft Dermis: Subjects with clinically significant pelvic organ prolapse Stage greater than or equal to 2, with surgical intervention using Axis device in the anterior, posterior, or combined (anterior and posterior) compartments.
Period: Overall Study
Arm/Group | Axis Allograft Dermis
Started | 74 (74 subjects were consented; however, 5 were screen failures and 1 did not receive the study device.)
Completed | 43
Not Completed | 31
Not completed — Lost to Follow-up | 17
Not completed — Moved out of state | 1
Not completed — Withdrawal by Subject | 7
Not completed — Screen failure | 5
Not completed — Did not receive study device | 1

BASELINE CHARACTERISTICS:
Groups:
- AXIS Allograft Dermis: Adult females with POP-Q Stage greater than or equal to 2 receiving AXIS Allograft Dermis for anterior, posterior or combined female pelvic floor repair.
Arm/Group | AXIS Allograft Dermis
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 74
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 27.9 (4.8)
Diabetes [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With POP-Q Stage Improvement Assessed by POP-Q Stage Improvement Based Upon Grading of Prolapse of the Anterior, Posterior, or Combined Anterior and Posterior Compartments Compared Between Baseline and One Year.
Description: The Pelvic Organ Prolapse Quantification system (POP-Q) is used to measure pelvic organ prolapse. POP-Q Stages are:
  Stage 0: No prolapse is demonstrated Stage 1: The criteria for stage 0 are not met, but the most distal portion of the prolapse is greater than 1 cm above the level of the hymen Stage 2: The most distal portion of the prolapse is greater than or equal to 1 centimeter proximal to or distal to the plane of the hymen Stage 3: The most distal portion of the prolapse is greater than 1 centimeter below the plan of the hymen but protrudes no further than 2 centimeters less that the total vaginal length in centimeters Stage 4: The distal portion of the prolapse protrudes to at least (TVL-2) centimeters.
  Improvement at one year is categorized as follows:
  Cured: Pop-Q Stage reduced to 0 or 1, or improved by 2 stages from baseline Improved: POP-Q Stage > 1, but improved by 1 stage from baseline Failed: POP-Q Stage stayed the same or increased in severity from baseline
Time Frame: 1 year
Population: Participants with clinically significant pelvic organ prolapse of Stage 2 or higher with surgical intervention using Axis Allograft Dermis in the anterior, posterior or combined (anterior and posterior) compartments.
Measure: Count of Participants; unit: Participants
Arm/Group | AXIS Allograft Dermis
Number analyzed (Participants) | 46
Participants
  Cured | 35
  Improved | 4
  Failed | 7

2. Secondary Outcome: Percentage of Participants With POP-Q Stage Improvement Assessed by POP-Q Stage Improvement Based Upon Grading of Prolapse of the Anterior, Posterior, or Combined Anterior and Posterior Compartments Compared Between Baseline and Six Weeks
Description: as for outcome 1
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AXIS Allograft Dermis
Number analyzed (Participants) | 65
Participants
  Cured | 63
  Improved | 1
  Failed | 1

3. Secondary Outcome: Percentage of Participants With POP-Q Stage Improvement After POP Repair With Axis Assessed by POP-Q Stage Improvement Based Upon Prolapse Grading of the Anterior, Posterior, or Combined Anterior and Posterior Compartments Between Baseline and Six Months
Description: as for outcome 1
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- AXIS Allograft Dermis: Adult females with POP-Q Stage greater than or equal to 2 receiving AXIS Allograft Dermis for anterior, posterior or combined female pelvic floor repair at 6 months
Arm/Group | AXIS Allograft Dermis
Number analyzed (Participants) | 57
Participants
  Cured | 46
  Improved | 5
  Failed | 6

4. Secondary Outcome: Percentage of Participants With POP-Q Stage Improvement Assessed by POP-Q Stage Improvement Based Upon Grading of Prolapse of the Anterior, Posterior, or Combined Anterior and Posterior Compartments Compared Between Baseline at 24 Months
Description: as for outcome 1
Time Frame: 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AXIS Allograft Dermis
Number analyzed (Participants) | 46
Participants
  Cured | 36
  Improved | 2
  Failed | 8

5. Secondary Outcome: Percentage of Participants With POP-Q Stage Improvement After POP Repair With Axis Assessed by POP-Q Stage Improvement Based Upon Prolapse Grading of the Anterior, Posterior, or Combined Anterior and Posterior Compartments Between Baseline at 36 Months
Description: as for outcome 1
Time Frame: 36 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AXIS Allograft Dermis
Number analyzed (Participants) | 43
Participants
  Cured | 27
  Improved | 7
  Failed | 9

6. Secondary Outcome: Change in Participant Sexual Satisfaction From Baseline After Pelvic Organ Prolapse Repair With Axis Allograft Dermis Measured by Participant Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) at 6 Months
Description: The PISQ-12 is the Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12). Sexual Function in women after pelvic organ prolapse repair with Axis Allograft Dermis measured by PISQ-12 at 6 months. The scores range from 0-48 with lower scores indicating better sexual function. Scores are calculated by totaling the scores for each question with (4) always, (3) usually, (2) sometimes, (1) seldom, and (0) never. Reverse scoring is used for items 1, 2, 3 and 4. The short form questionnaire can be used with up to two missing responses. To handle missing values, the sum is calculated by multiplying the number of items by the mean of the answered items.
Time Frame: Baseline and 6 months
Population: The 19 participants who completed the PISQ-12 at the 6 month follow up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Axis Allograft Dermis: Participants with clinically significant pelvic organ prolapse Stage greater than or equal to 2, with surgical intervention using Axis device in the anterior, posterior, or combined (anterior and posterior) compartments.
Arm/Group | Axis Allograft Dermis
Number analyzed (Participants) | 19
score on a scale
  6 months | -3.1 (10.4)
  Baseline | 16.8 (8.1)

7. Secondary Outcome: Change in Patient Sexual Satisfaction From Baseline After Pelvic Organ Prolapse Repair With Axis Allograft Dermis Measured by Participant Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) at 12 Months
Description: as for outcome 6
Time Frame: Baseline and 12 months
Population: The 17 participants who completed the PISQ-12 at the twelve month follow up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- AXIS Allograft Dermis: Participants with clinically significant pelvic organ prolapse of Stage 2 or higher with surgical intervention using Axis Allograft Dermis in the anterior and/or posterior compartment.
Arm/Group | AXIS Allograft Dermis
Number analyzed (Participants) | 17
score on a scale
  12 months | -2.9 (6.9)
  Baseline | 16.8 (8.1)

8. Secondary Outcome: Change in Patient Sexual Satisfaction From Baseline After Pelvic Organ Prolapse Repair With Axis Allograft Dermis Measured by Participant Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) at 24 Months
Description: as for outcome 6
Time Frame: Baseline and 24 months
Population: The 13 participants who completed the PISQ-12 at the 24 month follow up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AXIS Allograft Dermis
Number analyzed (Participants) | 13
score on a scale | -2.2 (5.1)

9. Secondary Outcome: Change in Patient Sexual Satisfaction From Baseline After Pelvic Organ Prolapse Repair With Axis Allograft Dermis Measured by Participant Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) at 36 Months
Description: as for outcome 6
Time Frame: Baseline and 36 months
Population: The 19 participants who completed the PISQ-12 at the 36 month follow up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AXIS Allograft Dermis
Number analyzed (Participants) | 19
score on a scale
  36 month | 11.9 (6.9)
  Baseline | 16.8 (8.1)

10. Secondary Outcome: Percentage of Participants Responding "Very Much Better" or "Much Better" on Patient Global Impression of Improvement for Urogenital Prolapse (PGI-I) at 12 Months
Description: The PGI-I Index consists of one question and was collected at 12 months. The question is "Check the box that best describes how your condition is now, compared with how it was before you had the operation." There are seven possible responses including, "very much better," "much better," "a little better," "no change," "a little worse," "much worse," and "very much worse and the subject chooses one response.
Time Frame: 12 months
Population: The 48 participants who completed the PGI-I at the 12 month follow up visit.
Measure: Number; unit: percentage of participants
Groups:
- Axis Allograft Dermis: Participants implanted with Axis Allograft Dermis who completed the PGI-I Questionnaire at 12 months.
Arm/Group | Axis Allograft Dermis
Number analyzed (Participants) | 48
percentage of participants | 87.5

11. Secondary Outcome: Percentage of Participants Responding "Very Much Better" or "Much Better" on Patient Global Impression of Improvement for Urogenital Prolapse (PGI-I) at 24 Months
Description: The PGI-I Index consists of one question and was collected at 24 months. The question is "Check the box that best describes how your condition is now, compared with how it was before you had the operation." There are seven possible responses including, "very much better," "much better," "a little better," "no change," "a little worse," "much worse," and "very much worse and the subject chooses one response.
Time Frame: 24 month
Population: The 46 participants who completed the PGI-I at the 24 month follow up visit.
Measure: Number; unit: percentage of participants
Groups:
- AXIS Allograft Dermis: The PGI-I Index consists on one question and was collected at 6 weeks. The question is "Check the box that best describes how your condition is now, compared with how it was before you had the operation." There are seven possible responses including "very much better," "much better," "a little better," "no change," "a little worse," "much worse" and "very much worse" and the subject chooses one response.
Arm/Group | AXIS Allograft Dermis
Number analyzed (Participants) | 46
percentage of participants | 87.0

12. Secondary Outcome: Percentage of Participants Responding "Very Much Better" or "Much Better" on Patient Global Impression of Improvement for Urogenital Prolapse (PGI-I) at 36 Months
Description: The PGI-I Index consists of one question and was collected at 36 months. The question is "Check the box that best describes how your condition is now, compared with how it was before you had the operation." There are seven possible responses including, "very much better," "much better," "a little better," "no change," "a little worse," "much worse," and "very much worse and the subject chooses one response.
Time Frame: 36 months
Population: The 42 participants who completed the PGI-I at the 36 month follow up visit.
Measure: Number; unit: percentage of participants
Groups:
- AXIS Allograft Dermis: Participants implanted with Axis Allograft Dermis
Arm/Group | AXIS Allograft Dermis
Number analyzed (Participants) | 42
percentage of participants | 88.1

13. Secondary Outcome: Change in Pelvic/Bladder Pain With Daily Activity Visual Analog Scale (VAS) Questionnaire From Baseline to 6 Weeks, 6 Months, 12 Months, 24 Months, 36 Months
Description: The Visual analog scales (VAS) Questionnaire is a questionnaire that asks the participant to mark a place on a scale that aligns with their level of pain. Participants were asked to make a vertical mark on a 10 centimeter line marked with "No Pain" and "Worst Pain" at each end and the line was measured to the tenths decimal place. A lower score indicates less pain.
Time Frame: Baseline and 6 weeks, 6 months, 12 months, 24 months, 36 months
Population: The participants who completed the VAS Questionnaire for Pelvic/Bladder Pain with Daily Activity at the 6 week, 6 month, 12 month, 24 month, and 36 month visits. Some participants either did not complete the questionnaire or did not complete it correctly and this accounts for the lesser total number of participant questionnaires analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AXIS Allograft Dermis
Number analyzed (Participants) | 61
units on a scale
  Baseline | 1.7 (2.6)
  6 week: number analyzed (Participants) | 58
  6 week | -.08 (2.4)
  6 month: number analyzed (Participants) | 52
  6 month | -1.0 (2.7)
  12 month: number analyzed (Participants) | 44
  12 month | -1.5 (2.8)
  24 month: number analyzed (Participants) | 42
  24 month | -1.1 (2.4)
  36 month: number analyzed (Participants) | 36
  36 month | 0.5 (1.6)

14. Secondary Outcome: Change in Pelvic/Bladder Pain With Sexual Activity Visual Analog Scale (VAS) Questionnaire From Baseline to 6 Weeks, 6 Months, 12 Months, 24 Months, 36 Months
Description: The Visual analog scales (VAS) Questionnaire is a questionnaire that asks the participant to mark a place on a scale that aligns with their level of pain. Participants were asked to make a vertical mark on a 10 centimeter line with the left end marker labeled "No Pain" and the right end marker labeled "Worst Pain." The line was measured to the tenths decimal place. Zero was the minimum value and 10 was the maximum value. Higher scores indicated a greater amount of pain.
Time Frame: Baseline and 6 weeks, 6 months, 1 year, 2 years, 3 years
Population: Participants who completed the VAS Questionnaire for Pelvic/Bladder Pain with Sexual Activity at the 6 week, 6 month, 12 month, 24 month, and 36 month visits. Some participants were not sexually active and this accounts for the lesser total number of participant questionnaires analyzed at certain visit intervals.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AXIS Allograft Dermis
Number analyzed (Participants) | 48
units on a scale
  Baseline | 1.8 (2.9)
  6 Week: number analyzed (Participants) | 35
  6 Week | -0.7 (2.9)
  6 Month: number analyzed (Participants) | 35
  6 Month | -0.3 (3.4)
  12 Month: number analyzed (Participants) | 33
  12 Month | -0.9 (2.9)
  24 Month: number analyzed (Participants) | 32
  24 Month | -1.0 (3.3)
  36 Month: number analyzed (Participants) | 28
  36 Month | -1.5 (3.3)

15. Secondary Outcome: Percentage of Participants Who Had Surgical Revision of the Index Prolapse Compartment(s) After Pelvic Organ Prolapse Repair With Axis
Description: Percentage of participants who had surgical revision of the index prolapse compartment(s) after pelvic organ prolapse repair with Axis from the time of the index procedure to the end of study visit.
Time Frame: 3 year
Population: The participants who had surgical revision of the index prolapse compartment(s) after pelvic organ prolapse repair with Axis from the time of the index procedure to the end of study visit.
Measure: Count of Participants; unit: Participants
Groups:
- AXIS Allograft Dermis: Participants with clinically significant pelvic organ prolapse of Stage 2 or higher with surgical intervention using Axis Allograft Dermis in the anterior, posterior or combined (anterior and posterior) compartments.
Arm/Group | AXIS Allograft Dermis
Number analyzed (Participants) | 68
Participants | 0

16. Secondary Outcome: Ratings for the Validated Surgical Satisfaction Questionnaire (SSQ-8) in Women Following Surgery to Correct Pelvic Organ Prolapse Repair With Axis Allograft Dermis at the 6 Week, 6 Month, 12 Month, 24 Month, and 36 Month Visits.
Description: The Surgical Satisfaction Questionnaire (SSQ-8) is a validated questionnaire consisting of eight questions assessing participant satisfaction with the results of their surgery to correct urinary incontinence and/or pelvic organ prolapse. Scoring is implemented with the mean average of the 8 scores multiplied by 25, yielding a potential range of scores from 0 to 100. The higher the score is, the greater the degree of surgical satisfaction.
Time Frame: 6 week, 6 month, 12 month, 24 month, and 36 month visits
Population: The subjects who completed the SSQ-8 Questionnaire at the 6 week, 6 month, 12 month, 24 month, and 36 month visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Axis Allograft Dermis
Number analyzed (Participants) | 65
score on a scale
  6 Weeks | 83.2 (15.9)
  Month 6: number analyzed (Participants) | 58
  Month 6 | 81.7 (20.2)
  Month 12: number analyzed (Participants) | 48
  Month 12 | 87.9 (13.8)
  Month 24: number analyzed (Participants) | 46
  Month 24 | 86.8 (14.8)
  Month 36: number analyzed (Participants) | 42
  Month 36 | 86.2 (17.3)

17. Secondary Outcome: Change in Pelvic Floor Distress Inventory (PFDI-20) Questionnaire After Pelvic Organ Prolapse Repair With Axis Allograft Dermis From Baseline to 6 Weeks, 6 Months, 12 Months, 24 Months, and 36 Months
Description: The Pelvic Floor Distress Inventory Questionnaire (PFDI-20) is a questionnaire with 20 questions that measures symptom distress and impact of health-related quality of life. The PFDI-20 has three scales:
  Pelvic Organ Prolapse Distress Inventory (POPDI-6), Colorectal-Anal Distress Inventory (CRADI-8), and Urinary Distress Inventory (UDI-6). Each of the 3 scales of the PFDI-20 is scored from 0 (least distress) to 100 (greatest distress). The sum of the scores of these 3 scales serves as the overall summary score of the PFDI-20 and ranges from 0 to 300. Higher scores indicate more distress.
Time Frame: Baseline and 6 weeks, 6 months, 12 Months, 24 Months, 36 Months
Population: Participants who completed the Pelvic Floor Distress Inventory (PFDI-20) Questionnaire at 6 week, 6 month, 12 Month, 24 Month, 36 Month visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AXIS Allograft Dermis
Number analyzed (Participants) | 60
score on a scale
  Baseline | 108.3 (59.6)
  6 Week: number analyzed (Participants) | 59
  6 Week | -58 (61.3)
  6 Month: number analyzed (Participants) | 51
  6 Month | -62.5 (63.4)
  12 Month: number analyzed (Participants) | 44
  12 Month | -69.4 (56.1)
  24 Month: number analyzed (Participants) | 42
  24 Month | -62.0 (63.6)
  36 Month: number analyzed (Participants) | 37
  36 Month | -62.7 (71.3)

18. Secondary Outcome: Change in the Participants Response on the Pelvic Floor Impact Questionnaire (PFIQ) From Baseline to 6 Weeks, 6 Months, 12 Months, 24 Months, 36 Months
Description: The Pelvic Floor Impact Questionnaire (PFIQ) measures impact of bladder, bowel, and vaginal symptoms on daily physical activity, travel, social/relationships, and emotional health. The PFIQ-7 has three scales: the Urinary Impact Questionnaire (UIQ-7), the Colorectal-Anal Impact Questionnaire (CRAIQ-7), and the Pelvic Organ Prolapse Impact Questionnaire (POPIQ-7). Response options range from 0 ("not at all") to 3 ("quite a bit"). Per scale, the mean score of answered items is multiplied by 33.3 to obtain the scale score (range 0-100) [4]. Summary scores are calculated by adding up the scale scores (range 0-300) [4]. Higher scores indicate more impact on daily activity.
Time Frame: Baseline and 6 weeks, 6 months, 12 Months, 24 Months, 36 Months
Population: Subjects who completed the Pelvic Floor Impact Questionnaire Questionnaire at 6 weeks, 6 month, 12 Month, 24 Month, and 36 Month visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AXIS Allograft Dermis
Number analyzed (Participants) | 60
score on a scale
  Baseline | 65.8 (63.4)
  6 Week: number analyzed (Participants) | 59
  6 Week | -31.5 (56.7)
  6 Month: number analyzed (Participants) | 51
  6 Month | -41.2 (66.5)
  12 Month: number analyzed (Participants) | 44
  12 Month | -46 (72.1)
  24 Month: number analyzed (Participants) | 42
  24 Month | -48.8 (65.9)
  36 Month: number analyzed (Participants) | 37
  36 Month | -44.9 (70.8)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the index procedure through study completion. Thus, the timeframe duration over which adverse events were collected is three years post index procedure.
Arm/Group | AXIS Allograft Dermis
All-Cause Mortality (participants affected / at risk) | 0/68
Serious Adverse Events (participants affected / at risk) | 1/68
Other Adverse Events (participants affected / at risk) | 7/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXIS Allograft Dermis (N=68)
Hematoma (Surgical and medical procedures) | 1 (1) — Retroperitoneal pelvic hematoma resulting in severe anemia, responded to 4 units of blood transfused.
Wound dehiscence (Surgical and medical procedures) | 1 (1) — Wound dehiscence with fever, bilateral abscess drained. Wound breakdown, repaired. Possible mechanical trauma caused both compartments wound breakdown.
Pelvic abscess. (Infections and infestations) | 1 (1) — Post-operative pelvic abscess. Drained by Interventional Radiology. No evidence of fistula.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXIS Allograft Dermis (N=68)
Pain (Lasting > 6 weeks post-operatively) (Surgical and medical procedures) | 3 (3) — Procedure related pelvic pain
Wound dehiscence (Skin and subcutaneous tissue disorders) | 4 (4) — One participant had a perineal separation. One participant had a superficial separation of incision. One participant had a 1 cm vaginal exposure. One participant had a vaginal posterior separation 1 x 2 cm.

LIMITATIONS AND CAVEATS:
The study N was small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-10-24): https://cdn.clinicaltrials.gov/large-docs/48/NCT01541748/Prot_SAP_000.pdf